CLINICAL TRIAL: NCT06585579
Title: ORIGYNE (MUCO232) - the Effect of Mucogyne® Ovule on Wound Healing
Brief Title: The Effect of Mucogyne® Ovule on Wound Healing (ORIGYNE)
Acronym: ORIGYNE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MUCO232; 2022-A02640-43 (Other: ID-RCB)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Cervicovaginitis

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mucogyne group (Experimental): For each eligible patient, the study will consist of:
  * A Screening/Inclusion visit
  * A treatment period (application of the medical device Mucogyne® ovule) for 21 days
  * An End Of Study visit (Day 21 (+10) after surgery)
  Interventions: Device: Mucogyne Ovule
- Control group (No Intervention): standard of care e.i no treatment

INTERVENTIONS:
Device: Mucogyne Ovule — In Mucogyne group, patient will receive 2 boxes of Mucogyne® ovule. 24 hours after intervention, the patient will apply Mucogyne® ovule, 1 ovule per day for 10 days, to be repeated as needed (for practices' homogenisation, after the 10th day, it is recommended to apply one ovule every second day, until EOS visit)
  Arms: Mucogyne group

SUMMARY:
This clinical investigation is a post-market clinical follow-up performed to confirm the performance and safety of the Mucogyne® ovule medical device in promoting the process of wound healing, when used in accordance with its approved labelling, in the context of local cervicovaginal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women who had undergone localized surgery (laser or loop electrosurgical excision procedure (LEEP) conization) for cervical or vaginal dysplasia,
2. Is able to understand the study related information and to give a written informed consent,
3. Has signed the informed consent form before beginning any study procedure,
4. Has no condition that may interfere with the study assessments,
5. Agrees not to use other vaginal products than those planned in the study protocol, during participation in the study,
6. Is able to comply with protocol requirements and respect the conditions of the study,
7. Affiliated to the Social Security system.

Exclusion Criteria:

1. Previous vaginal surgery within the year preceding the inclusion in the study,
2. Known hypersensitivity to any of the medical device ingredients,
3. Patient with local infectious lesions in the area to be repaired.
4. Patient who had used anti-inflammatory drugs (regular intake) or anticoagulants during the month preceding the inclusion in the study,
5. Patient who had a history of diseases known to disturb wound healing (e.g. systemic, heart, and renal diseases, coagulation disorders, immunedeficiency, connective tissue disorders, diabetes, anemia (with hemoglobin level < 9 g/dl) and hemophilia),
6. Immunosuppressive treatment,
7. Heavy cigarettes smoker (i.e., more than 15 cigarettes or equivalent/day, according to the patient and their documented records),
8. Patients under judicial protection or under guardianship and patients deprived of freedom,
9. Has any other severe chronic or acute medical or psychiatric condition that in the judgment of the Investigator, could interfere with the study assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To confirm the performance of Mucogyne® ovule in wound healing promotion | Day 0 to day 21(+10)
  The primary endpoint is a composite endpoint derived with the following criteria:
  * Inflammation evaluated with a 5-point scale (none, mild, moderate, severe, very severe) and not assessed,
  * Edema evaluated with a 5-point scale (none, mild, moderate, severe, very severe) and not assessed,
  * Abrasion evaluated with a 5-point scale (none, mild, moderate, severe, very severe) and not assessed,
  * Coalescence evaluated with a 3-point scale (none, partial, total) and not assessed.
  * Opening of the cervix (only for cervical wound) evaluated with a 4-point scale (closed, slightly open, open, gaping) and not assessed.

SECONDARY OUTCOMES:
To assess the aspect of the epithelium 3(+1) weeks after surgery | Day 0 to day 21(+10)
  Criteria assessing the aspect of the epithelium (such as presence of mucosa, stroma, presence and quality of mucus, opening of the cervix, presence or absence of inflammation, edema, vulvo-vaginal abrasions, coalescence, adherence, leucorrhoea and bleeding at contact)
To assess the performance of Mucogyne® ovule in symptoms relief | Day 0 to day 21(+10)
  Vaginal symptoms (dryness, itching, burning, discharge) will be assessed by the patient using a 4-point scale (1 = absent, 2 = mild, 3 = moderate, 4 = severe) at 3 (+1) weeks after surgery
To assess the performance of Mucogyne® ovule in reducing postoperative side effects and complications | Day 0 to day 21(+10)
  Postoperative side-effects (i.e. postoperative bleeding, infection and impairment of daily activities, etc.) will be assessed using a questionnaire. For the assessment of hemorrhage, the amounts of bleeding will be checked with a pictorial blood assessment chart.
To assess change in clinical status | Day 0 to day 21(+10)
  Change in clinical status will be assessed by the Investigator using Clinical Global Impressions scale, (CGI) at 3(+1) weeks after surgery
To assess compliance with the Medical Device use | Day 0 to day 21(+10)
  Compliance with the Medical Device use will be assessed by number of days of use
To assess the safety of Mucogyne® ovule | Day 0 to day 21(+10)
  Number, nature and characteristics of any incident reported: incidence, seriousness, severity, resolution

CONTACTS AND LOCATIONS:
Overall Officials: Oana BERNARD, MD, Study Director — Chief Scientific Officer
Locations (3):
- France (3):
  - CHU Amiens-Picardie, Amiens
  - CHU Besançon, Besançon
  - Hôpital Nord Franche-Comté, Trévenans